CLINICAL TRIAL: NCT03369002
Title: A Phase 1, Open Label, Non-Randomized Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Oral Seladelpar in Subjects With Varying Degrees of Hepatic Impairment and Healthy Matched Control Subjects With Normal Hepatic Function
Brief Title: Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Seladelpar in Subjects With Hepatic Impairment and Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CB8025-11732
Record Dates: First submitted 2017-11-16; First posted 2017-12-11 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment
MeSH Terms: interventions — seladelpar; (2-methyl-4-(5-methyl-2-(4-trifluoromethyl-phenyl)-2H-(1,2,3)triazol-4-ylmethylsulfanyl)phenoxy)acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Normal (Experimental): Child-Pugh Score: N/A
  Subjects will receive a single 10 mg oral dose of seladelpar
  Interventions: Drug: seladelpar
- Mild Impairment (Experimental): Child-Pugh Score: A (5 to 6 points)
  Subjects will receive a single 10 mg oral dose of seladelpar
  Interventions: Drug: seladelpar
- Moderate Impairment (Experimental): Child-Pugh Score: B (7 to 9 points)
  Subjects will receive a single 10 mg oral dose of seladelpar
  Interventions: Drug: seladelpar
- Severe Impairment (Experimental): Child-Pugh Score: C (10 to 15 points)
  Subjects will receive a single 10 mg oral dose of seladelpar
  Interventions: Drug: seladelpar

INTERVENTIONS:
Drug: seladelpar — Oral single dose 10 mg
  Other Names: MBX-8025

SUMMARY:
This Phase 1 open label study is being conducted to directly characterize the pharmacokinetic (PK) profiles of seladelpar following administration of a single oral dose in subjects with varying degrees of hepatic impairment (HI) compared to healthy matched control subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent (signed and dated) and any authorizations required by local law.
* Willing to be confined to CRU for the entire duration required by the protocol.
* Male or female, between 18 and 80 years of age.
* Healthy subject with normal liver function must be non-smoker and no use of other tobacco or nicotine-containing products. Subject with HI must be non-smoker, or smoke ≤10 cigarettes per day during the study.
* Healthy subject must not be taking any prescribed or non-prescribed medications unless permitted. Subject with HI will be allowed to take their chronic medications unless excluded by the protocol.

Exclusion Criteria:

* Pregnant or lactating women.
* Treatment with another investigational drug or device within 30 days prior to study drug administration.
* Has donated or lost a significant volume of blood within 56 days or plasma within 7 days prior to Check-in day.
* Inability to swallow medication.
* Positive test for drugs of abuse and/or positive alcohol test at Screening or Day -1.
* Positive test at Screening for HBsAg, hepatitis C virus (HCV), or HIV.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | 5 days
Time to reach maximum concentration (Tmax) | 5 days
Area under of the curve (AUC0-t and AUC0-∞) | 5 days
Elimination of half-life (t1/2) | 5 days
Apparent terminal elimination rate constant (λz) | 5 days
Total body clearance (CL/F) | 5 days
Volume of distribution (Vz/F) | 5 days

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - DaVita Clinical Research, Lakewood, Colorado
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota
  - Vrg & Noccr, Knoxville, Tennessee